CLINICAL TRIAL: NCT04962737
Title: Efficacy of Non-invasive Neuromodulation NESA Through Somatosensory Evoked Potentials and Sympathetic-cutaneous Responses in Healthy Subjects
Brief Title: Non-invasive Neuromodulation NESA Through Somatosensory Evoked Potentials and Sympathetic-cutaneous Responses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Principal Investigator, University of Las Palmas de Gran Canaria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NESAJaen
Record Dates: First submitted 2021-07-09; First posted 2021-07-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: physical therapy modality; Electric Stimulation Therapy; Evoked Potentials; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive Neuromodulation (Experimental): Non-invasive Neuromodulation Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Non-invasive Neuromodulation

INTERVENTIONS:
Device: Non-invasive Neuromodulation — The electrodes will be placed with the help of gloves and adapted socks for 1 hour, twice a week, until 10 intervention sessions are completed. In addition, depending on the session, an adhesive electrode will be placed at the level of C7. Characteristics of microcurrents: pulsed monophasic rectangular wave with a pulse of 1.3 s and pause of 300 ms, voltage 3 mV and intensity 0.5 μA.

SUMMARY:
Somatosensory evoked potentials are crucial in determining the physiological changes of potentials in nerve pathways. Although their main function is diagnostic, the investigators have recently been used as a physiological test to determine physioelectric changes in healthy subjects to study applied stimuli, such as laser, pain or electrotherapy.

DETAILED DESCRIPTION:
The general configuration of the study consists of a study before and after the block of sessions to be determined, and differences of all the variables measured before and after NESA therapy will be compared through the mechanisms of somatosensory evocations.

Given its potential use, the objective of this study is to determine if there are changes in the somatosensory evoked potentials of the ulnar, median, tibial, peroneal and vagus nerves when non-invasive neuromodulation NESA is applied, which is used as a physiotherapy treatment. for objectives such as pain, vegetative affectations and sleep disorders.

The variables of the study will be collected at two time points: before the intervention and at the end of the intervention.

The statistical analysis will be an intention-to-treat analysis. For the main outcomes variables a two factor ANOVA will-be performed (intervention-time) with a post-hoc analysis with kruskal wallis correction correction. Statistical significance will be defined as p <0.05

ELIGIBILITY:
Inclusion Criteria:

* Healthy people
* Optimal cognitive abilities and mentally competent to participate in the study.
* In condition to complete the study questionnaires.

Exclusion Criteria:

* Focal mononeuropathies in both upper and lower limbs
* Peripheral neuropathy.
* Patients with implanted functioning pacemakers / defibrillators. Patients with bleeding disorders. Patients being treated with anticoagulants. Patients on antiplatelet therapy.
* Present some of the contraindications for a treatment with NESA XSIGNAL®: pacemakers, internal bleeding, do not apply electrodes on skin in bad condition, with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and / or electricity phobia.
* Not having signed the informed consent.
* Present any injury or pathology during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Response speed of the central and peripheral nervous system to a stimulus 1 | Up to 1 month
  The Somatosensory Evoked Potentials of both median and ulnar nerves will be evaluated.
  Neurophysiological tests of the nervous system that functionally assesses the nerve pathways of the central and peripheral nervous system.
  For its evaluation, distal stimuli are generated in the wrists in the range of 3-4Hz with intensities above the sensitive threshold and below the pain threshold.

SECONDARY OUTCOMES:
Response speed of the central and peripheral nervous system to a stimulus 2 | Up to 1 month
  Somatosensory Evoked Potentials of both Posterior Tibial and Peroneal nerves will be evaluated.
  Neurophysiological tests of the nervous system that functionally assesses the nerve pathways of the central and peripheral nervous system.
  For its evaluation, distal stimuli are generated in the wrists in the range of 3-4Hz with intensities above the sensitive threshold and below the pain threshold.
Response speed of the central and peripheral nervous system to a stimulus 3 | Up to 1 month
  Somatosensory Evoked Potentials of the sensory auricular branch of the vagus nerves will be evaluated.
  Neurophysiological tests of the nervous system that functionally assesses the nerve pathways of the central and peripheral nervous system.
  Stimulations and recordings will be carried out only in the left auditory pavilion (since the right, due to the connection with the sinoatrial node of the heart by means of vagus efferences, can cause, according to the reports consulted, alteration of the heart rhythm and presyncope). Stimulations will be performed by means of a needle connected to the stimulator equipment, or in the tragus, by means of atrial surface electrode or auriculotherapy needle dipole.
Response speed to sensitive stimuli in the palms of the hand and sole of the feet | Up to 1 month
  Several simultaneous bilateral recordings after stimuli in the palms of the hand and sole of the feet above the sensory threshold in the limb contralateral to the recording, with a time between stimuli greater than one minute, to avoid habituation of the response.
  The latency of the first maximum deflection, in millivolts.

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez-Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria

REFERENCES:
- [Result] Cheshire WP, Freeman R, Gibbons CH, Cortelli P, Wenning GK, Hilz MJ, Spies JM, Lipp A, Sandroni P, Wada N, Mano A, Ah Kim H, Kimpinski K, Iodice V, Idiaquez J, Thaisetthawatkul P, Coon EA, Low PA, Singer W. Electrodiagnostic assessment of the autonomic nervous system: A consensus statement endorsed by the American Autonomic Society, American Academy of Neurology, and the International Federation of Clinical Neurophysiology. Clin Neurophysiol. 2021 Feb;132(2):666-682. doi: 10.1016/j.clinph.2020.11.024. Epub 2020 Dec 22. PMID 33419664
- [Result] Cruccu G, Aminoff MJ, Curio G, Guerit JM, Kakigi R, Mauguiere F, Rossini PM, Treede RD, Garcia-Larrea L. Recommendations for the clinical use of somatosensory-evoked potentials. Clin Neurophysiol. 2008 Aug;119(8):1705-1719. doi: 10.1016/j.clinph.2008.03.016. Epub 2008 May 16. PMID 18486546
- [Result] Fallgatter AJ, Neuhauser B, Herrmann MJ, Ehlis AC, Wagener A, Scheuerpflug P, Reiners K, Riederer P. Far field potentials from the brain stem after transcutaneous vagus nerve stimulation. J Neural Transm (Vienna). 2003 Dec;110(12):1437-43. doi: 10.1007/s00702-003-0087-6. Epub 2003 Jan 1. PMID 14666414
- [Result] Usami K, Kawai K, Sonoo M, Saito N. Scalp-recorded evoked potentials as a marker for afferent nerve impulse in clinical vagus nerve stimulation. Brain Stimul. 2013 Jul;6(4):615-23. doi: 10.1016/j.brs.2012.09.007. Epub 2012 Oct 11. PMID 23088852